CLINICAL TRIAL: NCT06340178
Title: CT-guided Lung Biopsy Risk Optimization Method - Effect of Fluid Application in the Pleural Cavity and the Gravitational Effect of Pleural Pressure
Brief Title: CT-guided Lung Biopsy Risk Optimization Method
Acronym: BROM-I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-00246
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pneumothorax; Biopsy, Needle; Risk Factors; Radiology, Interventional
Keywords: Image-Guided Biopsy; Risk Factors; Tomography; Biopsy; Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid administration (Experimental): Fluid is given in pleural or subpleural space during CT-guided lung biopsy.
  Interventions: Procedure: Fluid application during ct-guided lung biopsy
- No fluid administration (No Intervention): No additional fluid is given prior to the CT-guided lung biopsy.

INTERVENTIONS:
Procedure: Fluid application during ct-guided lung biopsy — Injection of a small amount of fluid (max. 20 ml sodium chlorid) in the pleural cavity at the biopsy site
  Arms: Fluid administration

SUMMARY:
The purpose of this randomized controlled study is to evaluate the extent to which injection of a small amount of fluid in the pleural cavity at the biopsy site may reduce the risk of pneumothoraces, in addition to patient positioning to allow biopsy in gravity-dependent areas of the lung.

DETAILED DESCRIPTION:
Study participants with written consent and the percutaneous, CT-guided lung biopsy already regularly indicated by the referring doctors (e.g., oncology) will be part of this study and will be randomized directly before the intervention. After randomization, the intervention is performed by Interventional Radiology, either with or without prior fluid administration into the pleural space. Three samples are taken using either an 18G or 20G coaxial needle, and any complications are treated according to the clinical standard. The lung biopsy will be only performed if clinically indicated and is not a study-specific intervention; data about the lung biopsy, like internal DICOM images of them retrieved from Inselspital's Picture Archiving and Communication System (PACS), laboratory results, and clinical information are retrieved from RIS (radiological information system) and iPDOS® and KISS by Epic® (electronic medical record) and the associated histopathological findings from the Institute of Pathology, University of Bern, will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent (knowledge of project languages), >18 years.
* Indeterminate or suspicious lung lesion unsuitable for transbronchial biopsy or Status after unsuccessful transbronchial biopsy
* Indication for biopsy given by referring specialist (in patients).

Exclusion Criteria:

* Preintervention bleeding into the pleural cavity
* More than 1 lesion should be biopsied at the same time
* Infiltration of the thoracic wall
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pneumothorax | Immediate after biopsy, expected to be on average 5 minutes
  Reduction of pneumothorax occurrence in patients with biopsy in dependent lung areas and pleural fluid administration compared to patients with biopsy in dependent lung areas without fluid administration. Immediately after the lung biopsy, the final CT scan of the intervention is used to check whether a pneumothorax is present or not - i.e. whether there is new air in the pleural cavity.

SECONDARY OUTCOMES:
Number of patients with bleeding | Immediate after biopsy, expected to be on average 5 minutes
  Local bleeding in lung parenchyma
Number of patients with chest tube placement | Immediate after biopsy, expected to be on average 5 minutes
  Chest tube placement if pneumothorax is more than 2 cm immediate after biopsy or progressive pneumothorax over time
Number of patients with air embolism | Immediate after biopsy, expected to be on average 5 minutes
  Evidence of air embolism in the postprocedural CT image

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brönnimann, MD, Principal Investigator — Department of Diagnostic, Interventional and Paediatric Radiology, Inselspital, Bern University Hospital, University of Bern, Freiburgstrasse 10, 3010 Bern, Switzerland;
Locations (1):
- Inselspital, Bern University Hospital, University of Bern, Freiburgstrasse 10, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data repository
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study closure
Access Criteria: Request to study P.I.